CLINICAL TRIAL: NCT03903549
Title: A Positron Emission Tomography (PET) Study to Investigate [18F]D6-FP-DTBZ ([18F]P17-059) for Potential Use as a Radioligand for Vesicular Monoamine Transporter (VMAT2)
Brief Title: Initial Investigation of [18F]P17-059 in Parkinson's Disease Patients and Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Five Eleven Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: JH-181698
Record Dates: First submitted 2019-04-03; First posted 2019-04-04 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brain uptake and kinetics in Parkinson patients (Experimental)
  Interventions: Drug: [18F]P17-059
- Brain uptake and kinetics in healthy volunteers (Experimental)
  Interventions: Drug: [18F]P17-059
- Dosimetry in healthy volunteers (Experimental)
  Interventions: Drug: [18F]P17-059

INTERVENTIONS:
Drug: [18F]P17-059 — Injection of < 10 mCi [18F]P17-059 followed by PET/CT scanning
  Other Names: [18F]D6FP; [18F]D6FPDTBZ

SUMMARY:
This study investigates the initial safety profile of [18F]P17-059 in healthy volunteers including dosimetry determination, and compares regional brain uptake and kinetics of [18F]P17-059 in Parkinson's disease patients with regional brain uptake and kinetics of [18F]P17-059 in healthy volunteers.

ELIGIBILITY:
* Inclusion criteria (Healthy Volunteers)

  1. Healthy non-smoking males and females, as determined by medical history, physical examination, vital signs, clinical laboratory tests, and an electrocardiogram.

     1.1 Male subjects and their child bearing potential partners must be willing to use a reliable method of birth control for the duration of the study.

     1.2 Female subjects who are of childbearing potential must agree to use an adequate method of contraception for the duration of the study.
  2. Between 45-85 years old, inclusive.
  3. BMI between 18-32 kg/m2 inclusive.
  4. Have clinical laboratory test results within the reference ranges for the population or results within acceptable deviations that are not considered by the investigator to be clinically significant.
  5. All subjects and their partners of childbearing potential must commit to use two methods of contraception, one of which must be a barrier method, from the time of screening and throughout the study and until follow-up.
  6. Less than 195 cm (6 feet and 5 inches) tall in order to accommodate the whole body scanning.
  7. Have sufficient venous access.
  8. Willing to give written informed consent and to comply with the study restrictions.
* Inclusion criteria (PD patients)

  1. Signed and dated written informed consent.
  2. Male or Female.
  3. Age 45-90.
  4. Diagnosis of clinically established idiopathic PD consistent with the Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease (PD) (Postuma, et al., 2014).
  5. BMI between 18-32 kg/m2 inclusive.
  6. Have clinical laboratory test results within the reference ranges for the population or results within acceptable deviations that are not considered by the investigator to be clinically significant.
  7. All subjects and their partners of childbearing potential must commit to use two methods of contraception, one of which must be a barrier method, from the time of screening and throughout the study and until follow-up.
  8. Less than 195 cm (6 feet and 5 inches) tall in order to accommodate the whole body scanning.
  9. Have sufficient venous access.
  10. Absence of an established clinical movement disorder diagnosis other than Parkinson's disease.
  11. Symptoms mild in intensity, this includes Hoehn & Yahr ≤ 2 (Exceptions are allowed for subjects who meet criteria for Hoehn & Yahr stage 2/5 due to early onset of postural instability and/or gait impairment out of proportion to his/her other Parkinson signs and symptoms);
  12. Montreal Cognitive Assessment (MoCA) score ≥ 22;
  13. Can tolerate imaging visit procedures
  14. Willing to give written informed consent and to comply with the study restrictions.
  15. Female patients must have had her last natural menstruation at least ≥24 months prior to the Screening Visit or have been surgically sterilized prior to the Screening Visit. Male patients must use two methods of contraception in combination if his female partner is of childbearing potential; OR have been surgically sterilized prior to the Screening Visit.
  16. In the opinion of the investigator based on medical history and physical examination, can safely tolerate tracer administration and the scanning procedures.
* exclusion criteria (Healthy volunteers)

  1. Are currently enrolled in or discontinued within the last 30 days from a clinical trial involving an investigational drug or device (other than the study drug) or are currently enrolled in any other type of medical research.
  2. Are currently experiencing neuropsychiatric illness or severe systemic disease based on history and physical exam.
  3. Have participated in other research protocols in the last year such that radiation exposure would exceed the annual limits.
  4. Pregnant or nursing women.
  5. History of head trauma with prolonged loss of consciousness (>10 minutes) or any neurological condition including stroke or seizure (excluding childhood febrile seizure).
  6. History or presence of any clinically relevant hematological, hepatic, respiratory, cardiovascular, renal, metabolic, endocrine, or CNS disease or other medical conditions that are not well controlled, may put the subject at risk, could interfere with the objectives of the study, or make the subject unsuitable for participation in the study for any other reason in the opinion of the principal investigator.
  7. Suffer from claustrophobia and would be unable to undergo MRI and PET scanning.
  8. Any confirmed significant allergic reactions against any drug, or multiple allergies.
  9. Currently uses prescription medications, over-the-counter drugs or herbal remedies such as St. Johns Wort) which cannot be discontinued 14 days (or < 5 half-lives, whichever is longer), prior to the PET scan and throughout the study. Exceptions include daily multiple vitamins.
* exclusion criteria (PD patients)

  1. Have a known CNS structural lesion such as stroke or tumor that likely accounts for their symptoms;
  2. Have current clinically significant cardiovascular disease or clinically important abnormalities on screening ECG (including but not limited to QTc > 450 msec);
  3. Are currently taking medications that are known to cause QT-prolongation;
  4. Are currently taking medications with narrow therapeutic windows (e.g. warfarin or other anticoagulant therapies);
  5. Are currently taking tetrabenazine (TBZ), valbenazine (Ingrezza), amphetamine type drugs;
  6. Has taken tetrabenazine (TBZ) in the preceding 3 months;
  7. Have a current clinically significant endocrine or metabolic disease, pulmonary, renal or hepatic impairment, or cancer (excluding localized basal cell carcinoma and in situ prostate cancer) that would interfere with completion of the study;
  8. Have a recent history (within the past year) of alcohol or substance abuse or dependence;
  9. Are females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable contraception. Females must not be pregnant (negative serum beta-hCG at the time of screening and negative urine beta-hCG on the day of imaging), must not be breastfeeding at screening, must avoid becoming pregnant and use adequate contraceptive methods for 14 days prior to and 24 hours after administration of 18F-D6-FPDTBZ for injection;
  10. Have had prior intracranial surgery; and
  11. Are receiving any investigational medications, or have participated in a trial with investigational medications within the last 30 days.
  12. Contraindications of MRI. Incidental findings on MRI scans that are pathognomonic for an active disease or pathological process which requires medical intervention will be exclusionary.
  13. History of, or suffers from, claustrophobia or feels that he or she will be unable to lie still on their back in the MRI or PET scanner.
  14. Urinary toxicology positive for nonprescribed substances
  15. Previous allergic reaction to the radiotracer ([18F]D6-FP-DTBZ) or substances of similar chemical structure or excipients.
  16. Diagnosis of secondary parkinsonism caused by a brain tumor, cranial trauma, or metabolic diseases (diabetes mellitus, hepatic insufficiency, alcoholism)

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Regional brain uptake of [18F]P17-057 in Parkinson patients compared healthy volunteers | 0 - 90 minutes post injection
  Quantitative estimates of [18F]P17-059 uptake in brain - SUV and non-displaceable Binding Potential
Cumulative organ [18F]P17-059 activity for estimates of radiation absorbed dose and effective dose | 0 - 240 minutes post injection
  Dosimetry

CONTACTS AND LOCATIONS:
Overall Officials: Martin Pomper, MD PhD, Principal Investigator — Johns Hopkins Medical School
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States